CLINICAL TRIAL: NCT04511104
Title: Effects of Exercise During the Acute Phase of Burns: A Multicenter Trial in Belgium
Brief Title: Effects of Exercise During the Acute Phase of Burns
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiteit Antwerpen (Other)
Collaborators: Research Foundation Flanders (Other)
Responsible Party: Principal Investigator, Ulrike Van Daele, University professor, Universiteit Antwerpen
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 11B8619N[BEL]
Record Dates: First submitted 2020-08-10; First posted 2020-08-12 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Burns
Keywords: Burns; Exercise rehabilitation; Exercise Therapy; Muscle wasting; Hypermetabolism; Insulin resistance
MeSH Terms: conditions — Burns; Muscular Atrophy; Insulin Resistance | interventions — Exercise; Standard of Care

STUDY DESIGN:
Intervention Model Description: Trial phase 1: All eligible subjects will be allocated to the intervention group until n=20 has been reached. To reduce staff workload during phase 1, patients will be allocated to the control group if staff capacity (max. 2 patients per full time employed physiotherapist) is saturated.
  Trial phase 2: When n=20 has been reached in the intervention group, all further eligible patients will be allocated to the control group for the remaining recruitment period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): Standard of care treatment:
  - including passive / assisted / active movements, stretching, functional exercise, scar treatment
  Duration: up to 8 weeks
  Interventions: Other: Standard of Care
- Exercise (Experimental): Standard of care + added exercises
  Exercise type: resistance and aerobic exercise
  Resistance Exercise: 3x / week (manual resistance, free weights, machines) Aerobic exercise: 2x / week (cycle ergometer, treadmill)
  Duration: up to 8 weeks
  Interventions: Other: Exercise; Other: Standard of Care

INTERVENTIONS:
Other: Exercise — Resistance and aerobic exercise in addition to standard of care rehabilitation
  Arms: Exercise
Other: Standard of Care — Standard of care rehabilitation

SUMMARY:
BACKGROUND:

Postburn changes in whole-body, glucose and protein metabolism are at their peak during the acute phase of severe burns. The resulting metabolic derangements lead to substantial muscle wasting, insulin resistance, which ultimately hampers full recovery and reintegration into society.

PURPOSE:

This quasi-experimental trial was initiated to investigate the effects of exercise-based rehabilitation on muscle wasting, insulin resistance, and quality of life during the acute phase of severe adult burns.

METHODS:

Moderate to severely burned adults (10-80%TBSA) will be recruited from two Belgian burn centres.

Subjects allocated to the intervention group will undergo an up to 8-week-long exercise program in addition to standard care rehabilitation. As part of the exercise program, participants will carry out progressive resistance and aerobic training, initiated as soon as medical safety and patient cooperation allow. Exercise type and dosage will be chosen according to patient status in terms of grafts, mobility, and strength.

The control group will receive standard care rehabilitation only, including passive, assisted, active range of motion exercise, functional exercise, and scar treatment.

The effect on muscle wasting will be determined by B-mode ultrasound-derived measures of quadriceps muscle layer thickness (QMLT) and rectus femoris cross sectional area, as well as peak force measurements by handheld dynamometry. Insulin resistance will be derived from the HOMA-2 index based on fasting plasma glucose and insulin. Quality of life will be determined by the EQ-5D-5L and Burn Specific Health Scale-Brief (BSHS-B) questionnaires.

The results of this clinical research will provide insight into the effects of exercise on both a fundamental and clinical spectrum.

DETAILED DESCRIPTION:
The added exercise intervention is initiated in line with the following readiness criteria, which will be checked prior to each training session:

Criteria:

* Mean arterial pressure (MAP) 60 - 110 mmHg
* Fraction of inspired oxygen (FiO2) <60%
* Partial pressure of oxygen / fraction of inspired oxygen (PaO2/FiO2) >200
* Respiratory rate <40 bpm
* Positive end expiratory pressure (PEEP) <10 cmH2O
* No high inotropic doses (Dopamine >10 mcg/kg/min or Nor/adrenaline <0,1 mcg/kg/min)
* Temp. 36 - 38,5°C
* Richmond Agitation Sedation Scale (RASS) -2 - +2
* Medical Doctor clearance
* Medical research council (MRC) score lower limbs ≥3

Accordingly, the post burn starting time differs per enrolled subject.

Exercises are administered as in-bed exercises or out-of-bed exercises, depending on whether subjects are able and allowed to engage in out-of-bed mobility.

Goal exercise intensity for resistance training is set at 60% peak force based on a weekly peak force measurement by hand-held dynamometry, or on a 3 RM in case of out of bed exercises. Goal aerobic exercise intensity is set at 50-75% peak Watts determined by a weekly cycle ergometer or treadmill ramp protocol.

ELIGIBILITY:
Inclusion Criteria:

* ≥10 - ≤80 %TBSA
* Burn depth: 2nd deep / 3rd degree

Exclusion Criteria:

* Electrical burn (except flash burns)
* Associated injury: fracture lower limb
* Diabetes Mellitus type 1
* Central neurological/neuromuscular disorders (interfering with assessment/exercise)
* Cognitive / psychological disorders (interfering with cooperation)
* Cardiopulmonary disease (interfering with exercise safety)
* Pregnancy
* Palliative care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-05-04 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in quadriceps muscle layer thickness (QMLT) | Baseline - Hospital discharge (max. 8 weeks)
  Method: B-mode ultrasound on the anterior aspect of the thigh. Technique: maximal and minimal pressure Location: measured at 1/2 and 2/3 of the distance between anterior superior iliac spine and the superior pole of the patella.
  Analysis: An average of 3 trials will be recorded and analyzed using dedicated software
Change in rectus femoris cross sectional area (RF-CSA) | Baseline - Hospital discharge (max. 8 weeks)
  Method: B-mode ultrasound on the anterior aspect of the thigh. Technique: minimal pressure. Location: measured at the most proximal distance where the entire muscle belly is still visible on the ultrasound image.
  Analysis: An average of 3 trials will be recorded and analyzed using dedicated software.

SECONDARY OUTCOMES:
Change in insulin resistance | Baseline - Hospital discharge (max. 8 weeks)
  Method: HOMA-2 calculated by fasting plasma glucose and insulin

OTHER OUTCOMES:
Change in isometric peak force (knee extension) | Baseline - Hospital discharge (max. 8 weeks)
  Method: Hand-held dynamometry (Lafayette instrument Co. Europe, U.K.). Isometric peak fore is measured by a 'make' manoeuvre with a fixation band disallowing movement.
  Test position: Supine with a fixation band fixed to the hospital bed. Analysis: Best of 3 trials
Change in isometric peak force (hip flexion) | Baseline - Hospital discharge (max. 8 weeks)
  Method: Hand-held dynamometry (Lafayette instrument Co. Europe, U.K.). Isometric peak fore is measured by a 'make' manoeuvre with a fixation band disallowing movement.
  Test position: Supine with a fixation band fixed to the hospital bed. Analysis: Best of 3 trials
Change in isometric peak force (hip extension) | Baseline - Hospital discharge (max. 8 weeks)
  Method: Hand-held dynamometry (Lafayette instrument Co. Europe, U.K.). Isometric peak fore is measured by a 'make' manoeuvre with a fixation band disallowing movement.
  Test position: Supine with a fixation band fixed to the hospital bed. Analysis: Best of 3 trials
Change in hand grip strength | Baseline - Hospital discharge (max. 8 weeks)
  Method: Baseline LITE hydraulic dynamometer Analysis: Best of 3 trials
Change in Burn Specific Health Scale-Brief (BSHS-B) | Baseline - Hospital discharge (max. 8 weeks)
  Burn-specific quality of life, measured by the Burn Specific Health Scale-Brief questionnaire (Dutch and French language version).
  Total score 152 (0 worst score, 152 best score), consisting of 6 subdomains:
  1) Body imagine (36 points) Simple abilities (36 points) Sexuality (24 points) Affect (32 points) Work (16 points) Interpersonal relationship (8 points)
Change in EQ-5D-5L | Baseline - Hospital discharge (max. 8 weeks)
  Overall quality of life, measured by EQ-5D-5L (Dutch and French language version) Total score: 25 points (0 worst score, 25 best score), consisting of 5 subdomains
  Mobility (5 points) Self-care (5 points) Usual activities (5 points) pain / discomfort (5 points) Anxiety / Depression (5 points) EQ overall health assessed on a Visual Analogue Scale, Total 0-100 (0 worst, 100 best score)
Number of adverse events | Baseline - Hospital discharge (max. 8 weeks)
  Recording of complications during exercise: Graft take, Wound infections, Medical, Cardio-respiratory safety

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Van Daele, Principal Investigator — University of Antwerp, Faculty of Medicine and Health Sciences
Locations (2):
- Belgium (2):
  - Ziekenhuis Netwerk Antwerpen Stuivenberg, Antwerp
  - Militaire Hospitaal Koningin Astrid, Neder-Over-Heembeek, Brussels

IPD SHARING:
Plan to Share IPD: No
Datasets will be made available upon request.